CLINICAL TRIAL: NCT02503072
Title: Variable Rewards Incentives for ART Adherence in Uganda
Brief Title: Rewarding Adherence Program - an Intervention Using Small Prizes Allocated by a Prize Drawing to Increase ARV Adherence
Acronym: RAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: Mildmay Uganda Limited (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1R34MH096609-01A1 (NIH)
Record Dates: First submitted 2015-07-14; First posted 2015-07-20 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: HIV
Keywords: ARV adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prizes conditional on adherence (Active Comparator): Participants in this group are eligible for a prize drawing if they come on their scheduled clinic day. They receive the intervention 'Behavioral: Small lottery prizes based on adherence'.
  Interventions: Behavioral: Small lottery prizes based on adherence
- Prizes conditional on clinic visits (Active Comparator): Participants in this group are eligible for a prize drawing if they show 95% adherence or higher based on their MEMS-cap measured adherence. They receive the intervention 'Behavioral: Small lottery prizes based on timely clinic visits'.
  Interventions: Behavioral: Small lottery prizes based on timely clinic visits

INTERVENTIONS:
Behavioral: Small lottery prizes based on adherence — Clients coming for clinic visits have their MEMS data extracted, and if they show 95% adherence or higher are eligible to draw a number (1-6) out of a closed bag without looking; if they draw a '6' they win a small prize.
  Arms: Prizes conditional on adherence
Behavioral: Small lottery prizes based on timely clinic visits — Clients coming for clinic visits have their patient booklet checked to confirm that they came on their scheduled day; if so, they are eligible to draw a number (1-6) out of a closed bag without looking; if they draw a '6' they win a small prize.
  Arms: Prizes conditional on clinic visits

SUMMARY:
The goal of this study is to identify ways for implementing small prizes allocated by a drawing to improve adherence to antiretroviral medication in an HIV clinic in Kampala, Uganda. The study is called Rewarding Adherence Program (RAP).

DETAILED DESCRIPTION:
The proposed 3-year study will develop and test RAP for incentivizing ART clients to remain engaged in care and highly adherent to their medication. Phase 1 of the project will consist of focus groups with patients, clinic providers and directors, and community leaders and will elicit information on barriers and facilitators of long-term retention and adherence maintenance, how to best implement the intervention to ensure acceptability and feasibility, and perceptions of the transportability of the planned intervention. Parameters of the intervention that will be probed include the frequency, type, and value of the prizes, and award presentation. Phase 2 will build on Phase 1 to develop and pilot test the RAP in a 20 months long randomized controlled trial (RCT) among clients who have been on ART for at least 2 years and have problems with missed clinic appointments or ART doses. Primary assessments will be administered at screening and months 4, 8, 14 and 20. In Phase 3 some adjustments to the intervention will be made after reviewing Phase 2 data, if needed, and then the intervention will be administered to the control group for 6 months to assess effects on adherence in this group (the original intervention group will not participate in this phase). Finally, the investigators will conduct focus groups with providers, implementers, and study participants to learn about implementation difficulties and areas for future improvement. Study findings will directly inform the design parameters of a larger, more rigorous evaluation in an R01 application that will focus on the cost-effectiveness and sustainability of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* patient at Mildmay Kampala clinic
* on antiretroviral medication (ARV) for at least two years
* shows recent adherence problems (missing a clinic visit or pharmacy refill in the last six months)

Exclusion Criteria:

* not able to understand study procedures and/or provide informed consent
* not fluent in either English or Luganda (the two main languages spoken around Kampala)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2013-03; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Medication Event Monitoring System (MEMS) cap measured adherence | 20 months
  Change in adherence over the course of the study
Medication Event Monitoring System (MEMS) cap measured adherence | 9 months
  Change in adherence over the first nine months of the study as an interim outcome

SECONDARY OUTCOMES:
Timely clinic visits | 20 months
  Number of timely clinic visits as a fraction of all scheduled clinic visits over the course of the study
Self-reported adherence | 20 months
  Adherence level as reported by the patient at month 20

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Linnemayr, PhD, Principal Investigator — RAND
Locations (1):
- Mildmay Uganda, Kampala, Uganda

REFERENCES:
- [Derived] Stecher C, Mukasa B, Linnemayr S. Uncovering a behavioral strategy for establishing new habits: Evidence from incentives for medication adherence in Uganda. J Health Econ. 2021 May;77:102443. doi: 10.1016/j.jhealeco.2021.102443. Epub 2021 Mar 16. PMID 33831632
- [Derived] Wagner GJ, Ghosh-Dastidar B, Mukasa B, Linnemayr S. Changes in ART Adherence Relate to Changes in depression as Well! Evidence for the Bi-directional Longitudinal Relationship Between Depression and ART Adherence from a Prospective Study of HIV Clients in Uganda. AIDS Behav. 2020 Jun;24(6):1816-1824. doi: 10.1007/s10461-019-02754-8. PMID 31813077
- [Derived] Linnemayr S, Stecher C, Mukasa B. Behavioral economic incentives to improve adherence to antiretroviral medication. AIDS. 2017 Mar 13;31(5):719-726. doi: 10.1097/QAD.0000000000001387. PMID 28225450